CLINICAL TRIAL: NCT02843490
Title: Correlation of Functional and Structural Outcomes With Serum Antibody Profiles in Patients With Neovascular Age-related Macular Degeneration Treated With Ranibizumab and Healthy Subjects: A Prospective, Controlled Monocenter Trial
Brief Title: Functional and Structural Outcomes in Neovascular Age-related Macular Degeneration
Acronym: CAPTAIN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johannes Gutenberg University Mainz (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Christina Korb, Dr. Med., Johannes Gutenberg University Mainz
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 469055
Record Dates: First submitted 2016-07-21; First posted 2016-07-25 (Estimated); Last update posted 2017-12-02 (Actual); Status verified 2017-11

CONDITIONS: Neovascular Age-related Macular Degeneration
Keywords: neovascular age-related macular edema; biomarker; ranibizumab; lucentis
MeSH Terms: interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ranibizumab treatment of nAMD patients (Experimental): nAMD patients will be treated with Ranibizumab (0.5 mg injection) 3 times within three months followed by individual therapy interval based on the clinical progress (PRN) up to 7 times. Analysis of specific biomarker.
  Interventions: Drug: Ranibizumab
- healthy subjects (No Intervention): Analysis of specific biomarker.

INTERVENTIONS:
Drug: Ranibizumab — Three injections (o.5 mg Ranibizumab) within the first three months is followed by an individual therapy interval based on the clinical progress (PRN)
  Other Names: Lucentis
  Arms: Ranibizumab treatment of nAMD patients

SUMMARY:
Several studies during the last years reported the involvement of anti-retinal autoantibodies in ocular disorders, such as AMD. These studies support the growing evidence of an immunological involvement in the pathogenesis of AMD. In the planned trial it is planned to enroll 70 subjects, i.e. 50 subjects with neovascular AMD and 20 healthy volunteers. The investigators will evaluate the change from Baseline (Visit 1) in BCVA score at Week 12 (visit 4) in the study eye of nAMD patients treated with Ranibizumab. Neovascular AMD patients (group 1) will be accompanied for 6 months and blood samples will be collected at baseline and monthly until Visit 7 for analysis of antibody profiles. Healthy volunteers (group 2) will be enrolled and a blood sample will be collected once for analysis of antibody profiles. Antibody profiles of all study participants will be analysed to address questions as defined in the outcome measures.

DETAILED DESCRIPTION:
Several studies during the last years reported the involvement of anti-retinal autoantibodies in ocular disorders, such as retinal vasculitis, retinopathy, retinitis pigmentosa and also AMD. These studies support the growing evidence of an immunological involvement in the pathogenesis of AMD. In the planned trial it is planned to enroll 70 subjects, i.e. 50 subjects with neovascular AMD and 20 healthy volunteers. The investigators will evaluate the change from Baseline (Visit 1) in BCVA score at Week 12 (visit 4) in the study eye of nAMD patients treated with Ranibizumab. AMD patients and healthy volunteers will be recruited at the Department of Ophthalmology of the University Medical Center, Johannes Gutenberg-University Mainz and included based on defined criteria. Neovascular AMD patients (group 1) will be accompanied for 6 months and blood samples will be collected at baseline and monthly until Visit 7 for analysis of antibody profiles. Ranibizumab is applied according to the manufacturer's recommendations and the "Stellungnahme der DOG, RG und BVA zu aktuellen therapeutischen Möglichkeiten bei der neovaskulären AMD" (December 2012). A loading dose of three injections within the first three months is followed by an individual therapy interval based on the clinical progress (PRN). Re-treatment after the upload of the three initial doses every 4 weeks will be performed in case of progression (PRN) based on the recommendations of the "Stellungnahme der DOG, RG und BVA zu aktuellen therapeutischen Möglichkeiten bei der neovasculären AMD" (December 2012). Healthy volunteers (group 2) will be enrolled and a blood sample will be collected once for analysis of antibody profiles.

Beside the analysis of primary endpoint, the investigators propose to analyze in detail the following questions:

Does the ranibizumab treatment have any effects on antibody profiles found in sera and do these changes correlate with the clinical course of the disease?

Additionally, the patient group can be divided into two subgroups: AMD patients with newly diagnosed neovascular AMD, who have not received anti-VEGF-treatment so far (naïve subjects) and AMD patients with neovascular AMD, who have not received any anti-VEGF treatment 3 months prior to inclusion in the study. This separation may help to answer the question if it is possible to differentiate between ranibizumab responder and non-responder with the help of antibody profiles.

ELIGIBILITY:
Inclusion Criteria (patients):

* Male or female
* Age ≥ 50 years
* Subfoveal, juxtafoveal and/or extrafoveal choroidal neovascularisation due to neovascular age-related macular degeneration in the study eye
* Visual acuity of 20/400 (ETDRS charts) or better in the study eye
* Ability of subject to understand character and individual consequences of clinical Trial
* Signed and dated informed consent of the subject must be available before start of any specific trial procedures
* Women with childbearing potential have to practice a medically accepted contraception during trial and a negative pregnancy test (urine) should be existent before trial. Reliable contraception are systematic contraceptives (oral, implant, injection) and diaphragm or condoms with spermicide. Women that are sterile by surgery or for more than two years postmenopausal can participate in the trial.

Inclusion Criteria (healthy subjects):

* Male or female
* Age ≥ 50 years

Exclusion Criteria (patients):

* Inability to obtain fluorescein angiography
* Ophthalmic Surgery or laser < 3 months before enrolment in one or both eyes
* Any history of intravitreal steroids in one or both eyes
* Systemic and/or intravitreal anti-VEGF-treatment < 3 months before enrolment in one or both eyes
* Patients with hypersensitivity against ranibizumab
* Ocular inflammation (including trace or above) or external ocular inflammation in the study eye
* Inability to give informed consent to participate in the study
* Pregnancy and lactation; Woman who are of childbearing age and not using medically acceptable effective contraception.
* Medical or psychological condition that would not permit completion of the trial or signing of informed consent (legal representative accepted)
* Participation in other clinical trials including an investigational drug or device during the present clinical trial or within the last 4 weeks.

Exclusion Criteria (Healthy subjects):

* Ophthalmic Surgery or laser < 3 months before enrolment
* Relevant eye diseases except age-related cataract in one or both eyes
* Inability to give informed consent to participate in the study
* Pregnancy and lactation; Woman who are of childbearing age and not using medically acceptable effective contraception.
* Medical or psychological condition that would not permit completion of the trial or signing of informed consent (legal representative accepted)
* Participation in other clinical trials including an investigational drug or device during the present clinical trial or within the last 4 weeks

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2016-08-05 (Actual); Primary Completion 2017-08-17 (Actual); Study Completion 2017-11-09 (Actual)

PRIMARY OUTCOMES:
Change in BCVA | Baseline - 12 weeks
  Change from Baseline (Visit 1) in BCVA score at Week 12 (visit 4) in the study eye.

SECONDARY OUTCOMES:
Change in BCVA | Baseline - 24 weeks
  Change from Baseline (Visit 1) in BCVA score at Week 24 (visit 7) in the study eye.
Change in retinal thickness | Baseline - 24 weeks
  Absolute change from baseline (Visit 1) in central retinal thickness, assessed by OCT at Week 24 (Visit 7) in the study eye.
Number of ranibizumab injections | 24 weeks
  Mean number of IVT ranibizumab injections needed up to Week 24 (Visit 7) in the study eye.

OTHER OUTCOMES:
Identification of biomarkers against retinal antigens | 24 weeks
  Identification of antibodies (biomarkers) against retinal antigens (anti cyclophilin B, heat shock protein (HSP) 10, HSP 70) in patients with neovascular AMD treated with ranibizumab and healthy subjects.
Validation of biomarkers | 24 weeks
  Validation of antibodies (biomarkers) against retinal antigens (anti cyclophilin B, heat shock protein (HSP) 10, HSP 70) in patients with neovascular AMD treated with ranibizumab and healthy subjects found in previous studies.
Correlation of functional and structural parameters | 24 weeks
  To correlate functional and structural parameters (BCVA and central retinal thickness) with the identified biomarkers to differentiate between initial and deferred responders.

CONTACTS AND LOCATIONS:
Overall Officials: Christina Korb, MD, Principal Investigator — Johannes Gutenberg-University Mainz, Germany
Locations (1):
- Clinical Trial Site, Department of Ophthalmology, University Medical Center Johannes Gutenberg University Mainz, Mainz, Germany

IPD SHARING:
Plan to Share IPD: No